CLINICAL TRIAL: NCT00113503
Title: A Multi-site Trial of Azathioprine Dosing in Crohn's Disease
Brief Title: Imuran Dosing in Crohn's Disease Study
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Insufficient enrollment
Sponsor: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Collaborators: Prometheus Laboratories (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: DK60083 (terminated); U01DK060083 (NIH)
Record Dates: First submitted 2005-06-08; First posted 2005-06-09 (Estimated); Last update posted 2017-10-06 (Actual); Status verified 2017-10

CONDITIONS: Crohn's Disease
Keywords: Inflammatory Bowel Disease, Crohn's disease, Crohn's Colitis
MeSH Terms: conditions — Crohn Disease; Inflammatory Bowel Diseases | interventions — Azathioprine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Azathioprine weight-based dose (Active Comparator)
  Interventions: Drug: Azathioprine weight-based dose
- Azathioprine individualised dose (Experimental)
  Interventions: Drug: Azathioprine individualised dose

INTERVENTIONS:
Drug: Azathioprine weight-based dose
  Other Names: Imuran
  Arms: Azathioprine weight-based dose
Drug: Azathioprine individualised dose
  Other Names: Imuran
  Arms: Azathioprine individualised dose

SUMMARY:
This study will compare two different dosing methods of azathioprine (IMURAN) in participants with Crohn's disease who are currently taking steroids (e.g. prednisone or budesonide)or who have just started steroids. The study can be up to 54 weeks long. All participants enrolled will receive active drug. Participants will take doses either based upon weight or based on the patient's ability to breakdown the drug (monitored by 6-thioguanine nucleotides (6-TGN) metabolite levels in the blood). All patients enrolled in the study will receive active study drug.

DETAILED DESCRIPTION:
This multi-center, double blind (patients and doctors do not know treatment group assignment), randomized (patients are put in 1 of 2 groups) clinical trial which will compare two 52-week-long azathioprine(AZA) dosing methods.

The patients enrolled will all be taking steroids (prednisone or budesonide)or have just been prescribed a steroid. The patients will be either in remission on steroids, but cannot taper off without a flare, patients who are on steroids and are still having Crohn's symptoms, or patients who need to start taking steroids.

After a two week screening period, patients fitting enrollment criteria will be begin taking study drug. Patients will begin to taper steroids per a set schedule, and taper off steroids completely by week 13. Patients who need to go back on steroids because of returned symptoms are allowed to, per a set schedule in the protocol. Patients will have monthly visits that include physical exams, blood tests and a quality of life questionnaire. Patients will be required to keep a diary of abdominal pain, liquid or soft stools and general well being.

After 6 months, only patients in remission (patients not on steroids, and not having active symptoms) will be allowed to continue for last 6 months of the study. Study visits during the last 6 months will be every 2 months, and include physical exams and blood tests, and a quality of life questionnaire.

Patients in the study may receive dose changes, and this will require additional blood tests for safety.

ELIGIBILITY:
Inclusion Criteria:

* 10-70 years-old., Weigh 20-100 kg (44-220 lbs).
* CD of the ileum, colon or ileocolon, verified by colonoscopy, barium enema, or small bowel series performed within 36 months
* Perianal fistulae will be eligible provided that the perianal disease does not account for the preponderance of symptoms.
* Have steroid-dependent, steroid-refractory or steroid naive CD.

  * Steroid-dependent CD: CDAI or mCDAI of < 150 while receiving prednisone 10-40 mg/day or budesonide 3-9 mg/day for at least 12 weeks prior to screening, but unable to taper prednisone below 10 mg/day or budesonide below 3 mg/day without experiencing a flare within the previous 6 months. Steroids must be at a stable dose for 2 weeks prior to screening (week #-2), prednisone at a dose of 10-40 mg/day and budesonide at a dose of 3-9 mg/day.
  * Steroid-refractory CD: currently moderately active CD (CDAI or mCDAI 200 - 450) despite treatment with 40 kg) or 0.5 mg/kg/day (if weighing 20 mg/day (if weighing prednisone <40 9 mg/day for the previous 4 weeks prior to the screening kg), or budesonide evaluation. Prednisone or budesonide must be at a stable dose for 2 weeks prior to screening (week #-2).
  * Steroid-naïve CD: currently moderately active CD, (CDAI or mCDAI 200 - 450) and one of the following:

    1. Despite treatment with aminosalicylates and/or antibiotics for the previous 4 weeks prior to the screening evaluation, who are candidates for prednisone or budesonide.
    2. Not currently on therapy, who are candidates for prednisone or budesonide
    3. Patients with prior exposure to steroids, who have not been treated with steroids for 4 weeks prior to screening, and are candidates for prednisone or budesonide Prednisone or budesonide will be started at the screening visit, at a dose of 40 mg/day or 9 mg/day and tapered per the steroid taper.

Patients who have started steroids up to 14 days prior to screening will also qualify as steroid naïve, however patient needs to be on 40 mg prednisone or 9 mg budesonide.

* Discontinue oral or rectal 5-Aminosalicylic acid (5-ASA) therapies, rectal steroids, ciprofloxacin or metronidazole at the screening visit.

Exclusion Criteria:

* CDAI > 450
* CD requiring hospitalization and intravenous (iv) corticosteroids, iv antibiotics or total parenteral nutrition (TPN).
* TPN or enteral nutrition of >1000 Calories/day (both TPN and elemental diets impact the CDAI).
* History of resection of more than 100 cm of small bowel, total proctocolectomy, or subtotal colectomy with ileorectal anastomosis
* Ileostomy or colostomy
* Severe fixed symptomatic stenosis of the small or large intestine
* Blood transfusion within 3 months before screening
* Treatment with 6-MP or AZA within the 6 months prior to screening
* Immunosuppressants or biologics 3 months before screening
* Treatment 2 weeks before screening:

  * Allopurinol;
  * Trimethoprim-sulfamethoxazole;
  * NSAIDs or aspirin >81mg/day;
  * Cholestyramine or other drugs interfering with enterohepatic circulation;
  * Furosemide and thiazide diuretics;
  * Fish-oil preparations.
* Discontinue use at screening: Oral or rectal 5-ASA, rectal steroids, metronidazole or quinolones
* Any prior treatment with natalizumab
* Presence of abnormal laboratory parameters:
* Carriage of hepatitis B surface antigen or positive hepatitis C antibody
* Lack of one acceptable form of contraception while receiving AZA
* Low TPMT activity

Ages: 10 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2005-07 (Actual); Primary Completion 2007-12 (Actual); Study Completion 2007-12 (Actual)

PRIMARY OUTCOMES:
Proportion of subjects achieving clinical remission at week #16. | 16 weeks
  For the steroid-dependent subjects, clinical remission was defined as complete withdrawal of corticosteroids, and Crohn's Disease Activity Index (CDAI) score <150 in adults, or modified CDAI (mCDAI) score <150 in children. For the steroid-refractory and the steroid-naıve subjects, clinical remission was defined as CDAI score <150 (or mCDAI <150 in children), and a reduction of at least 70 points from the baseline score (CDAI or mCDAI), and complete withdrawal of corticosteroids.

SECONDARY OUTCOMES:
Proportion of subjects maintaining clinical remission at week #28 | 28 weeks
Proportion of subjects maintaining clinical remission at week #52 | 52 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Stephen B Hanauer, MD, Principal Investigator — University of Chicago
Locations (15):
- United States (12):
  - Cedars-Sinai Medical Center, Los Angeles, California
  - Atlanta Gastroenterology Associates, LLC, Atlanta, Georgia
  - University of Chicago Pediatric Gastroenterology, Chicago, Illinois
  - University of Chicago, Chicago, Illinois
  - Johns Hopkins University, Baltimore, Maryland
  - Duluth Clinic, Duluth, Minnesota
  - Mayo Clinic, Rochester, Minnesota
  - Long Island Clinical Research Assoc., Great Neck, New York
  - Mt. Sinai Medical Center, New York, New York
  - University of North Carolina Chapel Hill, Chapel Hill, North Carolina
  - Cincinnati Children's Hospital, Cincinnati, Ohio
  - University of Pittsburgh, Pittsburgh, Pennsylvania
- Canada (3):
  - University of Alberta, Edmonton, Alberta
  - London Health Sciences Centre, London, Ontario
  - Hospital for Sick Children, Toronto, Ontario

REFERENCES:
- [Result] Dassopoulos T, Dubinsky MC, Bentsen JL, Martin CF, Galanko JA, Seidman EG, Sandler RS, Hanauer SB. Randomised clinical trial: individualised vs. weight-based dosing of azathioprine in Crohn's disease. Aliment Pharmacol Ther. 2014 Jan;39(2):163-75. doi: 10.1111/apt.12555. Epub 2013 Nov 17. PMID 24237037